CLINICAL TRIAL: NCT04787900
Title: Concurrent Validity and Reliability of the iPhone® Measurement Application to Evaluate Iliotibial Band Length
Brief Title: Reliability and Validity of iPhone Application for OBER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: KaratayUSonmezOber
Record Dates: First submitted 2021-03-04; First posted 2021-03-09 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-03

CONDITIONS: Reliability and Validity; Smartphone; Iliotibial Band Syndrome
MeSH Terms: conditions — Iliotibial Band Syndrome

STUDY DESIGN:
Intervention Model Description: wo experienced physiotherapists will evaluate the elasticity of both the dominant and non-dominant iliotibial bands after 2 minutes of warm-up before the evaluation. Measurements will be made by two physical therapists for each participant in different rooms without seeing each other. The examiners will carry out three measurements for both extremities, using both the bubble inclinometer and the iPhone® measurement app. A 5-minute passive rest will be give between measurements. All evaluations will be first conducted by Examiner 1 and then by Examiner 2. Measurement values will be record by a third physiotherapist. Data obtained from both devices will be compare in terms of validity and reliability using statistical analysis used in previous studies.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The Examiner 3 will be record the result by placing the device to be measured on the lateral projection of the midpoint of the femur. By preserving the participant's position, measurements will be make with the other device immediately and the values will bw record by the Examiner3.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iPhone measurement application (Experimental): For the measurement, the participant was asked to lie on his side and flex the knee to 90 degrees. The examiner stabilized the patient from the pelvis with one hand, and with the other hand brought the flexed leg of the participant to abduction and extension. The Examiner 3 recorded the result by placing the device to be measured on the lateral projection of the midpoint of the femur.
  Interventions: Device: iPhone measurement application
- Bubble inclinometer (Active Comparator): measurement will be done by the same method. For the measurement, the participant was asked to lie on his side and flex the knee to 90 degrees. The examiner stabilized the patient from the pelvis with one hand, and with the other hand brought the flexed leg of the participant to abduction and extension. The Examiner 3 recorded the result by placing the device to be measured on the lateral projection of the midpoint of the femur.
  Interventions: Device: Bubble inclinometer

INTERVENTIONS:
Device: iPhone measurement application — The iPhone measurement application will be used to ensure validity and reliability.
  Arms: iPhone measurement application
Device: Bubble inclinometer — Bubble inclinometer with proven validity and reliability will be used for this study.
  Arms: Bubble inclinometer

SUMMARY:
The validity and reliability of adduction angle measurement of hip with smartphone will be investigate.

DETAILED DESCRIPTION:
Our study is to investigate the intra-rater reliability, inter-rater reliability and concurrent validity of iPhone Measurement Applications to measure iliotibial band length in individuals without iliotibial band-related pathology. The aim of this study is to evaluate the intra-rater reliability, inter-rater reliability and concurrent validity of bubble inclinometer and iPhone Measurement Applications in the evaluation of iliotibial band tension in healthy individuals. This research is being done to determine if there are other more reliable, valid or innovative technological ways to measure iliotibial band length.

Participants:

A priori power analysis indicated that a minimum 16 or more participants should be enrolled the study for a correlation of 0.7, with an α level of .05 and power of 95%. The study protocol comply with the Declaration of Helsinki for Human Experimentation. Participants were excluded if they had hip or knee surgery in the past year and iliotibial band syndrome. All participants provide written informed consent. Permission for the study was obtained from KTO Karatay University Faculty of Medicine Drug and Non-Medical Device Research Ethics Committee with decision number 2019/012.

Two experienced physiotherapists will evaluate the elasticity of both the dominant and non-dominant iliotibial bands after 2 minutes of warm-up before the evaluation. Measurements will be made by two physical therapists for each participant in different rooms without seeing each other. The examiners will carry out three measurements for both extremities, using both the bubble inclinometer and the iPhone® measurement app. A 5-minute passive rest will be give between measurements. All evaluations will be first conducted by Examiner 1 and then by Examiner 2. Measurement values will be record by a third physiotherapist. Data obtained from both devices will be compare in terms of validity and reliability using statistical analysis used in previous studies.

All inclinometric measurements will be do by two independent blind examiners (B.S.U. and H.G.) and the range of motion (ROM) will be read directly from the devices by a third examiner.

Before the first measurement, the participant will be ask to warm up for five minutes. For the measurement, the participant will be ask to lie on his side and flex the knee to 90 degrees. The examiner will stabilize the patient from the pelvis with one hand, and with the other hand brought the flexed leg of the participant to abduction and extension. The Examiner 3 will be record the result by placing the device to be measured on the lateral projection of the midpoint of the femur. By preserving the participant's position, measurements will be make with the other device immediately and the values will bw record by the Examiner3.

After the first measurement, second and third measurements will be take at 2-minute passive intervals.

After the participants will complete their first examiner evaluation, they will move to the second examiner's room. The same protocol will be use for all measurements by the Examiner 2.

Instruments We will use 2 devices to measure iliotibial band length; bubble inclinometer (Baseline, Fabrication Enterprises Inc., New York) and iPhone® Measurement Applications (Apple Inc, California). The iPhone® Measurement Applications measurements will make with the iPhone 6s plus running IOS 13.3.1 (Apple Inc, California).

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 20 and 45 and agreed to participate the study.

Exclusion Criteria:

* Having hip or knee surgery

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-04-24 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
iPhone Measurement Application | 3 weeks
  Iliotibial band length of the participants will be measured with the iPhone Measurement Application

SECONDARY OUTCOMES:
Bubble inclinometer | 3 weeks
  Iliotibial band length of the participants will be measured with the Bubble inclinometer

CONTACTS AND LOCATIONS:
Locations (1):
- KTO Karatay University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No